CLINICAL TRIAL: NCT03020602
Title: A Phase I Study of BPM31510 Plus Vitamin K in Subjects With High-Grade Glioma That Has Recurred on a Bevacizumab Containing Regimen
Brief Title: BPM31510 in Treating Patients With Recurrent High-Grade Glioma Previously Treated With Bevacizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seema Nagpal (Other)
Responsible Party: Sponsor-Investigator, Seema Nagpal, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-38514; NCI-2016-01973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRN0035 (Other: Stanford Cancer Institute)
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Gliosarcoma; Recurrent Glioblastoma; Astrocytoma of Brain; Glioblastoma
MeSH Terms: conditions — Gliosarcoma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (BPM31510) (Experimental): Patients receive ubidecarenone injectable nanosuspension IV over 72 hours twice weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ubidecarenone Injectable Nanosuspension

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Ubidecarenone Injectable Nanosuspension — Given IV
  Other Names: BP31510; Coenzyme Q10 Injectable Nanosuspension; Ubiquinone Injectable Nanosuspension

SUMMARY:
This phase I trial studies the side effects and best dose of ubidecarenone injectable nanosuspension (BPM31510) in treating patients with high-grade glioma (anaplastic astrocytoma or glioblastoma) that has come back and have been previously treated with bevacizumab. BPM31510 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
Primary Objective:

* Assess the safety and tolerability of BPM31510 plus vitamin K in subjects with high-grade glioma(HGG), defined as anaplastic astrocytoma (AA) or glioblastoma (GB) that has recurred on a BEV containing regimen.

Secondary Objectives:

* To evaluate plasma pharmacokinetics (PK) when BPM31510 plus vitamin K is given to subjects with HGG recurrent on a BEV containing regimen.

Exploratory Objectives:

* Estimate the overall survival in subjects with HGG recurrent on a BEV containing regimen from the 1st day of infusion of BPM31510 plus vitamin K to death.
* To evaluate the effects of BPM31510 plus vitamin K on shifting HGG metabolism to aerobic respiration by PET imaging.
* To evaluate the effects of BPM1510 plus vitamin K on MRI imaging by Response Assessment in Neuro Oncology (RANO) criteria [specifically progression free survival (PFS) and response rate (RR)].
* To evaluate plasma pharmacodynamics (PD) when BPM31510 plus vitamin K is given to subjects with HGG recurrent on a BEV containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Have a life expectancy ≥ 6 weeks
* Have a Karnofsky Performance Score (KPS) ≥ 60
* Have pathologically proven GB, gliosarcoma (WHO IV), or anaplastic astrocytoma (WHO III) in recurrence after treatment with bevacizumab
* Be at least 14 days from the last administration of bevacizumab
* Be at least 28 days from last administration of cytotoxic chemotherapy or other investigational agent
* Have received radiation therapy with concurrent temozolomide. Total radiation dosage can range from 5400 to 6000 cGy administered in daily fractions of 150 to 200 cGy over 6 weeks, or the equivalent in a hypofractionated protocol (for example, 4000cGy in 15 fractions or 2500cGy in 5 fractions). Patients who are MGMT negative do not need to have received temozolomide.
* Have adequate organ and marrow function as follows (all required):

  * ANC ≥ 1500 mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 1.8 mg/dL or creatinine clearance > 50 mL/min Bilirubin ≤ 1.5 mg/dL
  * Alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
  * Aspartate transaminase (AST) ≤ 2.5 x ULN
  * Prothrombin time (PT) ≤ 1.5 x ULN
  * International Normalized Ratio (INR) ≤ 1.5 x ULN
  * Partial thromboplastin time (PTT) ≤ 1.5 x ULN
* Subjects of childbearing potential must agree to use hormonal or barrier birth control with spermicidal gel to avoid pregnancy during the study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Has a history of spontaneous or tumor related cerebral hemorrhage; or has cerebral hemorrhage as determined by the screening FDG PET CT and MRI. This does not include stable post operative blood products seen on a gradient echo MRI sequence.
* Has the any of the following cardiac history:

  * Active heart disease including myocardial infarction within previous 3 months
  * Symptomatic coronary artery disease
  * Arrhythmias not controlled by medication
  * Unstable angina pectoris
  * Uncontrolled or symptomatic congestive heart failure (NYHA class III and IV) 3.2.3 Uncontrolled or severe coagulopathies or a history of clinically significant bleeding within the past 6 months, including any of the following, but not limited to:
  * Epistaxis
  * Hemoptysis
  * Hematochezia
  * Hematuria
  * Gastrointestinal bleeding
  * Spontaneous or tumor related intracranial hemorrhage
* Known predisposition for bleeding such as von Willebrand's disease or other such condition(s)
* Uncontrolled concurrent illness that would limit compliance with study requirements, including any of the following, but limited to:

  * Uncontrolled infection.
  * Psychiatric illness/social situations
* Prior malignancy except for non melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 3 years prior to 1st dose of investigational drug
* Receiving any of the following medications:

  * Therapeutic doses of any anticoagulant, including low molecular weight heparin (LMWH). Concomitant use of warfarin, even at prophylactic doses, is prohibited
  * Digoxin, digitoxin, lanatoside C, or any type of digitalis alkaloids.
  * Colony stimulating factors (CSFs) that cannot be held during the monitoring period for dose limiting toxicities (DLT)
* Has significant toxicities from prior treatment that have not resolved or stabilized
* Known allergy to Coenzyme Q10
* Known allergy or adverse reaction to oral, subcutaneous, or intravenous vitamin K
* Is pregnant or lactating
* Known to be positive for the human immunodeficiency virus (HIV). Note: HIV testing is not required for eligibility, but if performed previously and was positive, the subject is ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with dose-limiting toxicities defined as thrombocytopenia >= grade 3, hemorrhage >= grade 3, and INR elevation >= grade 2 assessed by CTCAE v4.03 | Up to 28 days
  Will be tabulated at each dose, along with the result of the pooled adjacent violators algorithm as implemented in the Modified Toxicity Probability Interval (equal weights, and the weighted mean solver).

SECONDARY OUTCOMES:
Incidence of adverse events graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version (v)4.03 | Up to 30 days after last dose of BPM3150
  Will be tabulated separately for each dose cohort, by Medical Dictionary for Regulatory Activities (MedDRA) major organ system and severity.

OTHER OUTCOMES:
Brain tumor metabolism as measured by PET | Up to 8 weeks
  Standardized uptake value (SUV) of the HGG will be measured. SUV is the standard PET measure.
Overall survival (OS) | From the date of BPM31510 initiation to death, assessed for up to 3 years
  Kaplan-Meier survival estimates for OS will be presented for data at the maximum tolerated dose, with a 95% confidence interval using Greenwood's formula at 3.5 months and 7 months.
PFS assessed by RANO criteria | Up to 3 years
Response rate assessed by RANO criteria | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Seema Nagpal, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03020602/ICF_000.pdf